CLINICAL TRIAL: NCT01443260
Title: Phase I/II Study of Intraperitoneal Administration of GL-ONC1, a Genetically Modified Vaccinia Virus, in Patients With Peritoneal Carcinomatosis
Brief Title: A Study of GL-ONC1, an Oncolytic Vaccinia Virus, in Patients With Advanced Peritoneal Carcinomatosis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Genelux GmbH (Industry)
Responsible Party: Sponsor
Organization: Genelux Corporation (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Genelux - PO2; 2010-022680-35 (EudraCT Number)
Record Dates: First submitted 2011-09-20; First posted 2011-09-29 (Estimated); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Peritoneal Carcinomatosis
Keywords: oncolytic virus; oncolytic; GL-ONC1; Vaccinia; Vaccinia virus; Genelux; Genelux GmbH; peritoneal; peritoneal carcinomatosis; cancer; abdominal cancer; imaging
MeSH Terms: conditions — Peritoneal Neoplasms; Vaccinia; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: GL-ONC1 — A genetically-engineered vaccinia virus administered via intraperitoneal infusion through an indwelling catheter every 4 weeks for 4 cycles.

SUMMARY:
The purpose of this study is to determine whether GL-ONC1, an attenuated vaccinia virus, is safe when administered to patients with peritoneal carcinomatosis via an infusion within the abdominal cavity through an implanted catheter. The study seeks also to arrive at a recommended dose and schedule for future investigations, evidence of anti-tumor activity, detection of virus in body fluids, analysis of viral delivery to tumor and normal cells, and to evaluate if there is an antibody response to vaccinia virus.

DETAILED DESCRIPTION:
Peritoneal carcinomatosis includes a variety of tumors with extensive metastasis throughout the peritoneal cavity (inside surface of the abdomen) and can be found with gall bladder, liver, colon, appendix, ovarian, pancreas, mesothelioma, pseudomyxoma peritonei, rectal, small bowel and stomach cancers. It broadly includes multiple tumors that develop in and line the peritoneal abdominal cavity and linings. These tumors may be difficult to completely remove surgically and may recur despite conventional systemic chemotherapy, thereby resulting in poor patient outcomes. In preclinical studies, GL-ONC1, an oncolytic vaccinia virus, has shown the ability to preferentially locate, colonize and destroy tumor cells in more than 30 different human tumors. A Phase I clinical study focusing on the safety and tolerability of GL-ONC1 intravenously administered to patients with a variety of solid tumor entities has shown that GL-ONC1 is well-tolerated at therapeutic dose levels, with documented evidence of antitumor activity. This additional Phase I/II study seeks to evaluate GL-ONC1 administered repetitively every 4 weeks up to 4 cycles via infusion using an implanted catheter in the peritoneal cavity. In Phase I, patients will be individually assessed for safety and dose limiting toxicity. The study aims of Phase II portion are continued collection of safety information to better define the tolerability of GL-ONC1, as well as viral replication and the action or effect of GL-ONC1 in humans at the selected dose level and dosing schedule for future trials. Throughout both phases of the study, anti-tumor effects will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of histologically or cytologically documented, advanced stage of peritoneal carcinomatosis that is refractory to standard therapy, exhibiting a likely survival of > 4 months as being judged clinically.
2. Evidence of measurable disease.
3. Age ≥ 18 years.
4. ECOG (Eastern Cooperative Oncology Group Performance Status) ≤ 2.
5. Required baseline laboratory data include:

   * Absolute neutrophil count (ANC) ≥ 1.5 × 109/L.
   * Platelets ≥ 75 ×109/L
   * Haemoglobin ≥ 9.5 g/dL
   * Serum creatinine ≤ 2 × upper limit of normal(ULN)
   * Total Bilirubin ≤ 5 × ULN
   * AST/ALT ≤ 7.5 × ULN
   * Negative pregnancy test for females of childbearing potential
   * Serum albumin ≥ 2.5 g/dL.
   * If serum albumin level is < 2.5/dL,albumin substitution should take place until the threshold of ≥ 2.5 g/dL.
6. Willing and able to comply with scheduled visits, treatment plan, laboratory tests, implantation of the indwelling peritoneal catheter, as well as the respective drainage procedures.
7. All patients must agree to use highly effective contraception.

Exclusion Criteria:

1. Patients exhibiting objective evidence at baseline of brain metastases are excluded from participating.
2. Pregnant or breast-feeding women.
3. Primary tumors and metastases to tissues/organs which, under clinical judgment, will likely hinder survival for at least the next 4 months.
4. Patients with fever, any active immunosuppressive systemic infection or a suppressed immune system, including known HIV, as assessed within 14 days prior to study enrolment.
5. Concurrent vaccination or immunotherapy for 28 days before study therapy and during study treatment.
6. Patients on immunosuppressive therapy or with immune system disorders, including autoimmune diseases. Concurrent steroid use of not more than an equivalent of 20 mg/day prednisolone is allowed.
7. Prior splenectomy.
8. Previous organ transplantation.
9. Fully therapeutic coagulation therapy that does not allow the intraperitoneal insertion of a permanent catheter.
10. Patients with clinically significant dermatological disorders(e.g., eczema or psoriasis), any skin lesions or ulcers, any history of atopic dermatitis, or any history of Darier's disease (Keratosis Follicularis).
11. Clinically significant cardiac disease (New York Heart Association, Class III or IV: see Appendix 10)
12. Known allergy to ovalbumin or other egg products.
13. Concurrent use of antiviral agents active against vaccinia virus.
14. Prior gene therapy treatment or prior therapy with cytolytic virus of any type.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2012-02; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Determine safety of administering GL-ONC1 intraperitoneally by the evaluation of the number of patients experiencing Adverse Events (type, frequency, and severity) | Change from baseline over 24 hours, on days 2, 3, 4,5,6, 7 post treatment (Cycle 1) and change from baseline for Cycles 2- 4 CX/Days 1, 2, 3, 5, 8 post-treatment. Each cycle is 4 weeks and treatment will occur for a total of 4 cycles.
  The safety of GL-ONC1 will be assessed by the evaluation of the type, frequency, and severity of adverse events (AEs), changes in laboratory tests (haematological, chemistry, urinary), immunogenicity and physical examination

SECONDARY OUTCOMES:
Dose Level and Dose Schedule | End of Phase I (at 18 mo.), at monthly treatments, and after study completion (expected at 36 mo.)
  Determination of recommended dose and schedule for phase II portion of trial and future investigations by analysis of safety and efficacy data
Detection of Anti-tumor Activity | Tumor imaging [pre-study, mid-term (Day 43), after last treatment (Day 106), for 1 year @ 12-week intervals for patients with stable disease/better); Tumor markers and peritoneal cytologies collected on average over 4 months
  Sampling of evidence of anti-tumor activity via standard imaging practices, viral delivery to tumor and normal cells, and immune response activity.

CONTACTS AND LOCATIONS:
Overall Officials: Ulrich M. Lauer, Prof. Dr. med., Principal Investigator — University Hospital Tuebingen; Michael Bitzer, Prof.Dr.med., Principal Investigator — University Hospital Tuebingen
Locations (1):
- University Hospital Tuebingen, Tübingen, Germany

REFERENCES:
- [Derived] Lauer UM, Schell M, Beil J, Berchtold S, Koppenhofer U, Glatzle J, Konigsrainer A, Mohle R, Nann D, Fend F, Pfannenberg C, Bitzer M, Malek NP. Phase I Study of Oncolytic Vaccinia Virus GL-ONC1 in Patients with Peritoneal Carcinomatosis. Clin Cancer Res. 2018 Sep 15;24(18):4388-4398. doi: 10.1158/1078-0432.CCR-18-0244. Epub 2018 May 17. PMID 29773661
- See also: Click here for Related Information — https://genelux.com/clinical-publications/